CLINICAL TRIAL: NCT01320514
Title: A Randomized, Controlled Study to Evaluate Safety and Efficacy of Fibrin Sealant VH S/D 4 S-APR (Artiss) for Tissue Adherence and Hemostasis and To Improve Wound Healing in Subjects Undergoing Endoscopic Browlift
Brief Title: Efficacy and Safety of Fibrin Sealant (FS) VH S/D-APR for Hemostasis and Wound Healing in Endoscopic Browlift
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Nguyen, Davis B., M.D. (Individual)
Collaborators: Baxter BioScience (Industry)
Responsible Party: Davis B Nguyen, M.D., Davis B Nguyen, M.D.
Other Study IDs: Endoscopic Browlift
Record Dates: First submitted 2010-11-30; First posted 2011-03-22 (Estimated); Last update posted 2011-03-22 (Estimated); Status verified 2011-03

CONDITIONS: Compare Ecchymosis and Edema for Fibrin Sealant and no Fibrin Sealant
MeSH Terms: interventions — Fibrin Tissue Adhesive

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Fibrin Sealant (Artiss)
  Interventions: Drug: Fibrin Sealant (Artiss)

INTERVENTIONS:
Drug: Fibrin Sealant (Artiss)

SUMMARY:
The primary objective is to evaluate the safety and efficacy of Artiss (Fibrin Sealant) in reducing the incidence of early postoperative bruising and swelling.

ELIGIBILITY:
Inclusion Criteria:

* Subjects planned for endoscopic browlift, subjects who read, understand and sign the written informed consent, healthy female or male subjects, 18-75 years old, and subjects who are able and willing to comply with the protocal requirements

Exclusion Criteria:

* Subjects who had previous browlift, subjects indicated for concurrent facial surgeries, subjects considered to be active smokers, subjects with ecchymosis/edema on day 0, significant laboratory abnormalities, subjects with known bleeding or coagulation disorders, subjects treated with anti-coagulants.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects planned for endoscopic browlift; healthy female or male; age 18-75
Sampling Method: Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2010-12; Primary Completion 2011-05 (Estimated); Study Completion 2011-05 (Estimated)

PRIMARY OUTCOMES:
Comparison of ecchymosis and edema | 30 days

SECONDARY OUTCOMES:
Resolution of ecchymosis and edema, incidence of hematoma/seroma | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Davis B Nguyen, M.D., Principal Investigator — Davis B Nguyen, M.D.
Locations (1):
- Davis B Nguyen, M.D., Beverly Hills, California, United States